CLINICAL TRIAL: NCT01676727
Title: CoreValve® ADVANCE Direct Aortic Study
Brief Title: ADVANCE Direct Aortic Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Other Study IDs: Advance-DA
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-08

CONDITIONS: Aortic Stenosis; Valvular Heart Disease
Keywords: Transcatheter Aortic valve Implantation; Heart Valve Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CoreValve aortic valve: Implantation of CoreValve aortic valve via direct aortic approach
  Interventions: Device: CoreValve aortic valve

INTERVENTIONS:
Device: CoreValve aortic valve — Implantation of CoreValve aortic valve via direct aortic approach

SUMMARY:
This study is intended to collect data regarding the clinical utility, safety and performance of the Medtronic CoreValve® System for Transcatheter Aortic Valve Implantation (TAVI) in patients with severe symptomatic aortic valve stenosis for which treatment via direct aortic access (DA) is selected.

DETAILED DESCRIPTION:
This study is intended to collect data regarding the clinical utility, safety and performance of the Medtronic CoreValve® System for Transcatheter Aortic Valve Implantation (TAVI) in patients with severe symptomatic aortic valve stenosis for which treatment via direct aortic access (DA) is selected. As part of the study analysis, resource utilization together with the Quality of Life questionnaires data will provide an important input into cost effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Severe symptomatic aortic valve stenosis requiring treatment
2. Acceptable candidate for elective treatment with the Medtronic CoreValve® System according to the most recent version of the Medtronic CoreValve® Instructions For Use
3. 21 years of age or older
4. Patient is willing and able to comply with all protocol-specified follow-up evaluations
5. The patient or legal representative has been informed of the nature of the study and has consented to participate, and has authorized the collection and release of his/her medical information by signing a consent form ("Patient Informed Consent Form")
6. Patient will receive the CoreValve® device via direct aortic approach TAVI -

Exclusion Criteria:

1. Known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, clopidogrel, nitinol, or sensitivity to contrast media which cannot be adequately pre-medicated
2. Sepsis, including active endocarditis
3. Recent myocardial infarction (<30 days)
4. Left ventricular or atrial thrombus by echocardiography
5. Uncontrolled atrial fibrillation
6. Mitral or tricuspid valvular insufficiency (>grade II)
7. Previous aortic valve replacement (mechanical valve or stented bioprosthetic valve)
8. Evolutive or recent (within 6 months of implant procedure) cerebrovascular accident (CVA) or transient ischemic attack (TIA)
9. Patients with:

   1. Vascular conditions that make insertion and endovascular access to the aortic valve impossible, or
   2. Symptomatic carotid or vertebral arterial narrowing (>70%) disease, or
   3. Thoracic aortic aneurysm in the path of delivery system
10. Bleeding diathesis or coagulopathy
11. Patient refuses blood transfusion
12. Estimated life expectancy of less than 12 months unless TAVI is performed
13. Creatine clearance <20 mL/min
14. Active gastritis or peptic ulcer disease
15. Pregnancy or intent to become pregnant during study follow up
16. Patient is participating in another trial that may influence the results of this study

    -

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe aortic stenosis who are scheduled for an elective transcatheter aortic valve implantation and who are selected (e.g. because of an calcified femoral artery) to receive the CoreValve® device via direct aortic access.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Moat, M.D., Principal Investigator — The Royal Brompton Hospital; Giuseppe Bruschi, M.D., Principal Investigator — Azienda spedaliera Niguarda Ca' Granda Milano
Locations (9):
- Nemocnice Podlesi Trinec, Třinec, Czechia
- Hopital de Rangueil, Toulouse, France
- Universitätsklinikum Halle (Saale), Halle, Germany
- Italy (2):
  - Azienda spedaliera Spedali Civili Di Brescia, Brescia
  - Azienda spedaliera Niguarda Ca' Granda Milano, Milan
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven
  - Medisch centrum Leeuwarden, Leeuwarden
- United Kingdom (2):
  - Brighton and Sussex University Hospitals NHS Trust, Royal Sussex County Hospital, Brighton
  - Royal Brompton & Harefield NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled: All subjects enrolled in the trial
Period: Overall Study
Arm/Group | All Enrolled
Started | 100
Implanted | 92
Completed | 68
Not Completed | 32
Not completed — Death | 18
Not completed — Withdrawal by Subject | 6
Not completed — Screening failure | 5
Not completed — Not willing to attend 1-year visit | 2
Not completed — Valve explanted | 1

BASELINE CHARACTERISTICS:
Population: All enrolled population.
Arm/Group | All Enrolled
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.9 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 52
Region of Enrollment [Number; unit: participants]
  Czech Republic | 20
  Netherlands | 18
  United Kingdom | 7
  Italy | 33
  France | 15
  Germany | 7

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Description: Kaplan-Meier estimate of 30-day all-cause mortality.
Time Frame: 30 days post-implant
Population: all subjects who underwent an attempted implant of whom all were implanted with the CoreValve device via the direct aortic approach
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Implanted Population: All subjects who were implanted with the CoreValve.
Arm/Group | Implanted Population
Number analyzed (Participants) | 92
Percentage of subjects | 4.4 [1.4 to 10.0]

2. Secondary Outcome: Kaplan-Meier Estimate of Major Adverse Cardiovascular and Cerebrovascular Events (MACCE)
Description: The combined safety endpoint is defined as a composite of:
  * All-cause mortality
  * All stroke
  * Life-threatening bleeding
  * Acute kidney injury-Stage 3 (including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complication
  * Valve-related dysfunction requiring repeat procedure (BAV, TAVR, or SAVR)
  * High degree AV block requiring permanent pacemaker implantation
Time Frame: 1, 6 and 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Implanted Population
Number analyzed (Participants) | 92
Percentage of subjects
  1 month | 7.6 [3.4 to 14.2]
  6 months | 17.6 [10.6 to 26.1]
  12 months | 19.9 [11.7 to 29.6]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 1 year post-implant procedure.
Groups:
- Implanted Population: all subjects who underwent an attempted implant of whom all were implanted with the CoreValve device via the direct aortic approach
Arm/Group | Implanted Population
All-Cause Mortality (participants affected / at risk) | 16/92
Serious Adverse Events (participants affected / at risk) | 72/92
Other Adverse Events (participants affected / at risk) | 68/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanted Population (N=92)
Stroke-TIA (Vascular disorders) | 3 (3)
Bleeding (Vascular disorders) | 24 (34)
Myocardial Infarction (Cardiac disorders) | 1 (2)
Renal Failure (Renal and urinary disorders) | 12 (12)
New or worsened conduction disturbances and arrhythmias without pacemaker implant (Cardiac disorders) | 11 (13)
Permanent Pacemaker Implantation (Surgical and medical procedures) | 13 (13)
Vascular access site and access-related complications (Injury, poisoning and procedural complications) | 15 (17)
Failure of current therapy for AS requiring hospitalization or worsening congestive heart failure (Cardiac disorders) | 10 (13)
Sternotomy or thoracotomy related event (Surgical and medical procedures) | 2 (4)
(General disorders) | 55 (103) — Adverse events not associated with the use of the study device were collected without a specific adverse event term
(Cardiac disorders) | 3 (3) — Adverse events not associated with the use of the study device were collected without a specific adverse event term
(Infections and infestations) | 2 (2) — Adverse events not associated with the use of the study device were collected without a specific adverse event term
(Injury, poisoning and procedural complications) | 1 (1) — Adverse events not associated with the use of the study device were collected without a specific adverse event term
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanted Population (N=92)
(Injury, poisoning and procedural complications) | 1 (1) — Adverse events not associated with the use of the study device were collected without a specific adverse event term
(Cardiac disorders) | 31 (38) — Adverse events not associated with the use of the study device were collected without a specific adverse event term
(General disorders) | 51 (93) — Adverse events not associated with the use of the study device were collected without a specific adverse event term
(Product Issues) | 1 (1) — Adverse events not associated with the use of the study device were collected without a specific adverse event term
(Renal and urinary disorders) | 10 (11) — Adverse events not associated with the use of the study device were collected without a specific adverse event term
(Infections and infestations) | 1 (1) — Adverse events not associated with the use of the study device were collected without a specific adverse event term
(Surgical and medical procedures) | 4 (4) — Adverse events not associated with the use of the study device were collected without a specific adverse event term
(Vascular disorders) | 14 (15) — Adverse events not associated with the use of the study device were collected without a specific adverse event term

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less